CLINICAL TRIAL: NCT06478108
Title: Interventional Software IRSW-MIM Guided Immunotherapy for Advanced Solid Tumors: a Phase II Clinical Trial.
Brief Title: Interventional Software for Multi-immunotherapy of Solid Tumors
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Immuno (Guangzhou) Biomedicine S&T Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-IRSW-MIM-024
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Liver Cancer; Solid Tumor, Adult
Keywords: Solid Tumor; Medical device; Software; Immunotherapy; Interventional radiology
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRSW-MIM (Experimental)
  Interventions: Device: IRSW-MIM

INTERVENTIONS:
Device: IRSW-MIM — IRSW-MIM collects patient's data and outputs a therapeutical strategy for treating advanced solid tumors.

SUMMARY:
This trial is designed to investigate the safety, response rates and survival outcomes of patients with advanced solid tumors by intra-tumor (IT) injection of multiple drugs including CTLA4, PD1, and/or PDL1 antibodies combined with drugs-eluting beads loaded with IL2, chemodrug, anti-angiogenesis drug, et. al that will be recommended by an AI-based medical software named IRSW-MIM developed by a cooperating company.

DETAILED DESCRIPTION:
Malignant solid tumors including lung and liver cancers are the most common malignancy worldwide, and their mortality rates are very high. China has a huge population base with about 4,000,000 new cancer cases each year. More than 60% of the solid tumors in China are diagnosed at mid-to-late stage and have lost the chance of surgery. Recently a lot of therapeutic strategies have been developed and applied to clinic including targeted therapy and immunotherapy, but the overall therapeutic efficiency is still low. It is very difficult to treat patients with recurrent/refractory/metastatic advanced solid cancers and more alternative therapies are urgently needed.

Antibodies against CTLA4, PD1 and PDL1 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions. CTLA4 antibody ipilimumab has been widely effectively using to combine with PD1 or PDL1 antibody or other drugs, therefore, an AI-based medical software has been developed to help to determine the detailed combinations and dosages according to personalized medical condition such as sex, body weight, key organ functions, tumor types and their PDL1 level, status of MSI and TMB, previous treatment, et. al. This software, named interventional radiology appliable software for muti-immunothepy (IRSW-MIM), will be assessed by clinical applications on cancer patients.

This phase II clinical trial is to test the the safety, efficacy and survival benefit of the IRSW-MIM guided immunotherapy for advanced solid tumors, including PFS, ORR, DCT, and median survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of cancer.
2. Signed informed consent before recruiting.
3. Age above 18 years with estimated survival over 3 months.
4. Child-Pugh class A or B/Child score > 7; ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Birth control.
9. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance.

   Any contraindications for hepatic arterial infusion procedure:

   A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Allergic to contrast agent;
8. Any agents which could affect the absorption or pharmacokinetics of the study drugs
9. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the reccommended treatment generated by the medical device | 5 years
  Safety will be assessed by recording all types of advise effects upon and after the treatment.
Progression-free survival | 5 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Disease control rate | 5 years
  Disease control rate will be defined as objective response rate + steady disease rate.
Duration of remission (DOR) | 5 years
  DOR will be defined as the duration of the cancer remission

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China